CLINICAL TRIAL: NCT02315586
Title: Characterization of Apolipoprotein A-I Pathways in Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150017; 15-H-0017
Record Dates: First submitted 2014-12-11; First posted 2014-12-12 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Apoliprotein A-1; Natural History
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Participants will be enrolled at the NIH Clinical Center.
- 2: IPF subjects will be recruited from the INOVA Fairfax Advanced Lung Disease Program

SUMMARY:
Background:

- Idiopathic pulmonary fibrosis (IPF) is a chronic lung disease that becomes worse over time. There is currently no effective treatment for it. Researchers want to study the disease and learn new ways to treat it.

Objectives:

- To discover new pathways that are involved in pulmonary fibrosis. To develop new drugs that may be used to treat pulmonary fibrosis.

Eligibility:

* People at least 18 years old with IPF.
* Healthy volunteers at least 18 years old.

Design:

* Participants will be screened with medical history, questionnaire, and physical exam. They will have blood, lung, and walking tests and chest scans.
* All participants will have 1 study visit, including:
* Medical history and physical exam.
* Questions about their breathing.
* Blood tests.
* Breathing tests.
* Six-minute walk test.
* Pregnancy test.
* Chest x-ray (healthy volunteers) or chest CT scan (people with pulmonary fibrosis ).
* Small area of skin may be removed.
* Genetic tests of blood and skin samples. Participants will probably not be informed of any findings. Samples may be used to make stem cells for use in research. Participants may be contacted in the future to give consent for this research.
* Some participants will have repeat visits over many years, repeating many of the study tests.

DETAILED DESCRIPTION:
Idiopathic Pulmonary Fibrosis (IPF) is a chronic progressive disease that occurs primarily in older individuals, 55 to 75 years of age, with a median survival of approximately 3 years from time of diagnosis. At present, there are no effective treatments for patients with IPF. Levels of apolipoprotein A-I (apoA-I) have been found to be reduced in the lungs of patients with IPF, while administration of human apoA-I has been shown to reduce bleomycin-induced collagen deposition in a murine model. Here, we would like to assess whether apoA-I pathways modify lung cell biology in patients with IPF. This is a specimen procurement, clinical phenotyping and genotyping protocol that will assess whether holo-apoA-I and apolipoprotein A-I mimetic peptides, can attenuate key pathogenic manifestations of IPF, such as proliferation and extracellular matrix generation by pulmonary fibroblasts, which may serve as evidence to support future human clinical trials of apoA-I for the treatment of IPF. Furthermore, the identification of new apoA-I responsive genes and pathways that mediate fibroblast proliferation in IPF may provide insights into disease pathogenesis and identify new therapeutic targets. Lastly, if induced pluripotent stem (iPS) cells can be successfully shown to model responsiveness of lung cells to apoA-I therapy, then this approach may be expanded with the goal of providing a personalized medicine analysis that could in the future guide selection of the most effective therapy for individual patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patient:

Males and females over the age of 18 with a diagnosis of IPF.

EXCLUSION CRITERIA:

Patient:

Female subjects who are pregnant or lactating

INCLUSION CRITERIA:

Normal Volunteer:

Males and females over the age of 18 without IPF.

EXCLUSION CRITERIA:

Normal Volunteer:

Female subjects who are pregnant or lactating

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled at the NIH Clinical Center. IPF subjects will be recruited from the INOVA Fairfax Advanced Lung Disease Program and study procedures will be performed in the outpatient unit/day hospital at the NIH Clinical Center.@@@
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Specimen procurement, clinical phenotyping and genotyping that will assess whether holo-apoA-I and apolipoprotein A-I mimetic peptides, can attenuate key pathogenic manifestations of IPF | 5 years
  Therefore, we request participation of a maximum of 500 subjects (250 IPF patients and 250 non-IPF subjects) to ensure that we have a sufficient number of samples to achieve the goals of the study.

SECONDARY OUTCOMES:
The effects of stimulating cultures of primary pulmonary fibroblasts from IPF patients and subjects without IPF with apolipoprotein A-I will also be compared to the effects seen following stimulation with apolipoprotein E | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stewart J Levine, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0017.html